CLINICAL TRIAL: NCT05936879
Title: Effects of IMT ON Dyspnea, PF and Quality of Life in Patients With CABG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0308
Record Dates: First submitted 2023-06-14; First posted 2023-07-10 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Exercise
Keywords: functional capacity; lung capacity; rehabilitation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomized control trial in which two groups one is intervention and the other is controlled group .Patient in the Intervention group will be treated with routine pysical therapy, Inspiratory muscle training and early ambulation after surgery, whereas patients in the control group will be not be treated with these interventions and will rather undergo routine physical therapy (ankle pumps, hand pumps isometrics of upper and lower limbs).
  Patients in the intervention group will receive treatment until discharge from hospital.
Who Masked: Participant
Masking Description: A randomized control trial in which two groups one is intervention and the other is controlled group .Patient in the Intervention group will be treated with routine pysical therapy, Inspiratory muscle training and early ambulation after surgery, whereas patients in the control group will be not be treated with these interventions and will rather undergo routine physical therapy (ankle pumps, hand pumps isometrics of upper and lower limbs).
  Patients in the intervention group will receive treatment until discharge from hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training and early ambulation (Experimental): Intervention group will be treated with Inspiratory muscle training once in a week for at least 3 weeks
  Interventions: Other: Inspiratory muscle training
- physical therapy including ankle pumps, hand pumps isometrics of upper and lower limbs. (Experimental): Control group routine physical therapy including ankle pumps, hand pumps isometrics of upper and lower limbs once in a week for at least 3 weeks
  Interventions: Other: physical therapy including ankle pumps, hand pumps isometrics of upper and lower limbs.

INTERVENTIONS:
Other: Inspiratory muscle training — Group A: Intervention group will be treated with Inspiratory muscle training and early ambulation and routine physical therapy including ankle pumps,hand pumps isometrics of upper and lower limbs after surgery
  Arms: Inspiratory muscle training and early ambulation
Other: physical therapy including ankle pumps, hand pumps isometrics of upper and lower limbs. — Group B: Control group routine physical therapy including ankle pumps, hand pumps isometrics of upper and lower limbs
  Arms: physical therapy including ankle pumps, hand pumps isometrics of upper and lower limbs.

SUMMARY:
Patient in the Intervention group will be treated with routine pysical therapy, Inspiratory muscle training and early ambulation after surgery, whereas patients in the control group will be not be treated with these interventions and will rather undergo routine physical therapy (ankle pumps, hand pumps isometrics of upper and lower limbs).

Patients in the intervention group will receive treatment until discharge from hospital.

DETAILED DESCRIPTION:
A randomized control trial in which two groups one is intervention and the other is controlled group .Patient in the Intervention group will be treated with routine pysical therapy, Inspiratory muscle training and early ambulation after surgery, whereas patients in the control group will be not be treated with these interventions and will rather undergo routine physical therapy (ankle pumps, hand pumps isometrics of upper and lower limbs).

Patients in the intervention group will receive treatment until discharge from hospital. On the day of discharge they will be assessed using 6 minute walk test, Borg rate of perceive exertion and health related quality of life scale. Data will be analyzed using SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Both Gender patients
* Patients who agreed to participate
* Age: 35 to 55

Exclusion Criteria:

* Patients with history of Angioplasty or CABG
* Chronic Renal failure
* Cardiac arrhythmias
* History of stroke
* Unstable angina

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
6 Min walk test | 4 weeks
  The 6 min walk test is a sub-maximal exercise test used to assess aerobic capacity and endurance.It is also use to monitor your response to treatments for heart lung and other health problems.Provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.

SECONDARY OUTCOMES:
Spirometer: | 4 weeks
  A spirometer is used to measure pulmonary function test including FVC, FEV1 and FEV1/FVC ratio. The normal values of FEV1/FVC ratio are >0.70 and FVC, FEV1 are >80% of predicted age

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Faisal, MS.CPPT, Principal Investigator — Riphah International University
Locations (1):
- National hospital Lahore., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinheiro AR, Christofoletti G. Motor physical therapy in hospitalized patients in an intensive care unit: a systematic review. Rev Bras Ter Intensiva. 2012 Jun;24(2):188-96. English, Portuguese. PMID 23917769
- [Background] Shakouri SK, Salekzamani Y, Taghizadieh A, Sabbagh-Jadid H, Soleymani J, Sahebi L, Sahebi R. Effect of respiratory rehabilitation before open cardiac surgery on respiratory function: a randomized clinical trial. J Cardiovasc Thorac Res. 2015;7(1):13-7. doi: 10.15171/jcvtr.2015.03. Epub 2015 Mar 29. PMID 25859310
- [Background] Oliveira EK, Silva VZ, Turquetto AL. Relationship on walk test and pulmonary function tests with the length of hospitalization in cardiac surgery patients. Rev Bras Cir Cardiovasc. 2009 Oct-Dec;24(4):478-84. doi: 10.1590/s0102-76382009000500008. English, Portuguese. PMID 20305920
- [Background] Caso G, Vosswinkel JA, Garlick PJ, Barry MK, Bilfinger TV, McNurlan MA. Altered protein metabolism following coronary artery bypass graft (CABG) surgery. Clin Sci (Lond). 2008 Feb;114(4):339-46. doi: 10.1042/CS20070278. PMID 17953516